CLINICAL TRIAL: NCT01802684
Title: OPTIMOX-aflibercept as First-line Therapy in 49 Patients With Unresectable Metastatic Colorectal Cancer. A GERCOR Feasibility Single-arm Phase II Study.
Brief Title: OPTIMOX-aflibercept as First-line Therapy in Patients With Unresectable Metastatic Colorectal Cancer
Acronym: VELVET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VELVET C12-1; 2012-003521-25 (EudraCT Number)
Record Dates: First submitted 2013-02-26; First posted 2013-03-01 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Unresectable Metastatic Colorectal Cancer
Keywords: unresectable; metastatic; colorectal; cancer; OPTIMOX; aflibercept
MeSH Terms: conditions — Neoplasm Metastasis; Neoplasms | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OPTIMOX-aflibercept (Experimental): Induction therapy (sequence #1)
  * Regimen : aflibercept + modified FOLFOX7
  * Duration : 6 cycles (3 months) Maintenance after induction (sequence #2) First phase (sequence #2A)
  * Regimen : aflibercept + fluoropyrimidine (simplifed LV5FU2 or capecitabine)
  * Duration : 6 cycles (3 months) Second phase (sequence #2B)
  * Regimen : aflibercept +/- fluoropyrimidine (simplifed LV5FU2 or capecitabine) according to eligibility criteria for chemotherapy-free interval)
  * Duration : until PD or limiting toxicity Reintroduction (sequence #3)
  * Regimen : aflibercept + modified FOLFOX7
  * Duration : 6 cycles (3 months) Maintenance after reintroduction (sequence #4)
  * Regimen : aflibercept + fluoropyrimidine
  * Duration : until PD or limiting toxicity
  Interventions: Biological: aflibercept

INTERVENTIONS:
Biological: aflibercept — Aflibercept (VEGF Trap) Recombinant human protein, at 25 mg/ml Dose : 4 mg/Kg -Day 1, q2w Route of administration: Intravenous (60 min infusion)

SUMMARY:
Evaluation of feasibility of adding aflibercept to an oxaliplatin-based regimen rather than a continuous administration of chemotherapy until progression, in order to decrease the risk of severe toxicities.

DETAILED DESCRIPTION:
The addition of aflibercept to the standard FOLFIRI regimen as second-line therapy was evaluated in a large phase III study (EFC10262-VELOUR). This new combination significantly improved both PFS (4.7 to 6.9 months, HR=0.76; P=.00007) and OS (12.1 to 13.5 months, HR=0.82; P=.0032). In the evaluable population (86.5%), the tumor response rate was also improved when adding aflibercept (ORR=19.8% [16.4-23.2]) to the FOLFIRI regimen (ORR=11.1% [8.5-13.8]).

This trial will evaluate the feasibility of adding aflibercept to an oxaliplatin-based regimen as a first-line therapy , using the OPTIMOX strategy rather than a continuous administration of chemotherapy until progression, in order to decrease the risk of severe toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent, and willing and able to comply with protocol requirements,
2. Histologically proven adenocarcinoma of the colon and/or rectum,
3. Metastatic disease confirmed,
4. No prior therapy for metastatic disease (in case of previous adjuvant therapy, interval from end of chemotherapy to relapse must be >6 months for fluoropyrimidine alone or >12 months for oxaliplatin-based, bevacizumab-based, cetuximab-based therapy,
5. Duly documented inoperable metastatic disease, ie not suitable for complete carcinological surgical resection,
6. At least one measurable or evaluable lesion as assessed by CT-scan or MRI (Magnetic Resonance Imaging) according to RECIST v1.1,
7. Age ≥18 years,
8. ECOG Performance status (PS) 0-2,
9. Hematological status: neutrophils (ANC) ≥1.5x109/L; platelets ≥100x109/L; haemoglobin ≥9g/dL,
10. Adequate renal function: serum creatinine level <150µM,
11. Adequate liver function: serum bilirubin ≤3 x upper normal limit (ULN), alkaline phosphatase <5xULN,
12. Proteinuria <2+ (dipstick urinalysis) or ≤1g/24hour,
13. Baseline evaluations: clinical and blood evaluations performed no more than 2 weeks (14 days) prior to confirmation of eligibility, tumor assessment (chest X ray, CT-scan or MRI, evaluation of non-measurable lesions) no more than 3 weeks (21 days) prior to confirmation of eligibility,
14. For female patients of childbearing potential, negative serum or urine pregnancy test within 1 week (7 days) prior of starting study treatment,
15. Female patients of childbearing potential must commit to using reliable and effective methods of contraception during the trial and until at least six months after the end of study treatment. Females are neither pregnant nor in breastfeeding. Male patients with a partner of childbearing potential must agree to use effective contraception in addition to the contraceptive method used by their partner during the trial and until at least six months after the end of study treatment.
16. Registration in a national health care system (CMU included for France).

Exclusion Criteria:

1. History or evidence upon physical examination of CNS metastasis unless adequately treated (e.g. non irradiated CNS metastasis, seizure not controlled with standard medical therapy),
2. Exclusive bone metastasis,
3. Uncontrolled hypercalcemia,
4. Pre-existing permanent neuropathy (NCI grade ≥2),
5. Uncontrolled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg despite optimal medical therapy), or history of hypertensive crisis, or hypertensive encephalopathy,
6. Concomitant unplanned antitumor therapy (e.g. chemotherapy, molecular targeted therapy, immunotherapy/ radio-immunotherapy),
7. Treatment with any other investigational medicinal product within 28 days prior to study entry,
8. Other serious and uncontrolled non-malignant disease,
9. Other concomitant or previous malignancy, except: i/ adequately treated in-situ carcinoma of the uterine cervix, ii/ basal or squamous cell carcinoma of the skin, iii/ cancer in complete remission for >5 years,
10. Any other serious and uncontrolled non-malignant disease, major surgery or traumatic injury within the last 28 days
11. Patients with known allergy to any excipient to study drugs,
12. History of myocardial infarction and/or stroke within 6 months prior to study entry,
13. Bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Progression free survival at 6 months | time interval from inclusion to the date of first documented disease progression or death from any cause, whichever occurs first. Assessed at 6 months.

SECONDARY OUTCOMES:
Median Progression Free Survival | time interval from inclusion to the date of first documented disease progression or death from any cause, whichever occurs first. Assessed up to 3 years after the beginning of the study
duration of disease control (DDC) | sum of PFS of each active treatment course. Assessed up to 3 years after the beginning of the study
  DDC excludes:
  * Intervals between disease progression and re-initiation of treatment,
  * PFS of inactive treatment if PD occurs at first evaluation after treatment re-initiation
Overall Survival | time interval from inclusion to the date of death from any cause. Assessed up to 3 years after the beginning of the study.
tumor Response Rate (RR) | Assessed every 2 months during treatment period (- Estimated treatment duration per patient : 16 months).
  assessed using RECIST version 1.1 per sequence of therapy.
Health related Quality of life | Assessed from study entry to 1 month after last study drug administration and up to 3 years after the beginning of the study.
  EORTC QLQ C-30
Safety | Assessed from study entry to 1 month after last study drug administration, assessed up to 3 years after the beginning of the study
  The study will take into account all adverse events observed during and after drug administration, with a particular interest for:
  * Any AE
  * Any AE related to study treatment
  * Any serious AE
  * Any serious AE related to study treatment
  * Any NCI-CTC grade 3 or 4 AE
  * Any NCI-CTC grade 3 or 4 AE related to study treatment
  * Any AE causing discontinuation of study treatment
  * Any AE causing discontinuation of selected treatment only
  * Any AE related to study treatment causing discontinuation
  * Any AE causing a dose reduction of study medication
  * Any AE leading to death
  * Any AE related to study treatment leading to death.
Curative salvage surgery | assessed up to 3 years after the beginning of the study
  The number of patient with R0 and R1 curative salvage surgery will be assessed globally and per sequence of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Benoist Chibaudel, MD, Principal Investigator — Hôpital Saint Antoine
Locations (8):
- France (8):
  - Polyclinique de Bordeaux Nord, Bordeaux
  - Hôpital Henri Mondor, Créteil
  - CHU Dupuytren, Limoges
  - Hôpital Privé Jean Mermoz, Lyon
  - CH Mont de Marsan, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Institut Mutualiste Montsouris, Paris